CLINICAL TRIAL: NCT00001160
Title: Studies on Thyroid Nodules and Thyroid Cancer
Brief Title: Studies on Tumors of the Thyroid
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 770096; 77-DK-0096
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-25

CONDITIONS: Hurthle Cell Thyroid Cancer; Tall Cell Variant Thyroid Cancer; Follicular Thyroid Cancer; Thyroid Cancer; Papillary Thyroid Cancer
Keywords: Thyroid Fine Needle Biopsy; Radioiodine; Dosimetry; Natural History
MeSH Terms: conditions — Thyroid cancer, Hurthle cell; Adenocarcinoma, Follicular; Thyroid Neoplasms; Thyroid Cancer, Papillary | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thyroid cancer: Patients with thyroid cancer
  Interventions: Drug: 68-Gallium Dotatate
- thyroid nodules: Patients with thyroid nodules
  Interventions: Drug: 68-Gallium Dotatate

INTERVENTIONS:
Drug: 68-Gallium Dotatate — For evaluation risk/benefit evaluation

SUMMARY:
Participants in this study will be patients diagnosed with or suspected to have a thyroid nodule or thyroid cancer.

The main purpose of this study is to further understand the methods for the diagnosis and treatment of thyroid nodules and thyroid cancer. Many of the test performed are in the context of standard medical care that is offered to all patients with thyroid nodules or thyroid cancer. Other tests are performed for research purposes. In addition, blood and tissue samples will be taken for research and genetic studies.

DETAILED DESCRIPTION:
The purpose of this study is to gain knowledge and experience in the diagnosis and therapy of thyroid cancer using established best standard of care and new techniques and approaches as they are developed. Study subjects will include adults and children with thyroid nodules requiring diagnostic imaging and fine needle aspiration biopsy, surgery, radioiodine scanning or therapy, appropriate follow up, consisting of tumor markers monitoring and anatomical and functional imaging. The limitations and significance of serum thyroglobulin (Tg) measurement for diagnosing tumor recurrence will be assessed. The study will permit a continued evaluation of the risk/benefit ratio of already established methods of administering radioiodine therapy, including the impact of pre-treatment dosimetric calculations, individualizing treatment with radioiodine. Under this protocol, samples of benign nodules and cancer tissue specimens for research studies will be collected. Data and samples collected during routine clinical care will be used to address research questions utilizing a number of approaches including microscopy, immunohistochemistry, proteomics and molecular analysis. All research studies will relate to the diagnosis, natural history and therapy of thyroid tumors, regulation of thyroid function, and the effects of thyroid function on the body. Blood and urine specimens will be collected for research studies in both the hypothyroid and euthyroid state.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, adults or children >= 6 months+.
2. Patients with known or suspected thyroid nodules and/or thyroid cancer.
3. At risk family members of patients who have a genetic susceptibility to developing thyroid cancer.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Serious underlying medical conditions that restrict diagnostic testing or therapy such as renal failure, congestive cardiac failure or active coexisting non-thyroid carcinoma requiring intervention before thyroid cancer is addressed.

Ages: 6 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only those with thyroid nodules and/or thyroid cancer will be allowed to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1977-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of thyroid cancer | As clinically indicated
  Blood draws, CT and other scans, physical exams, surgery (if applicable), thyroid biopsy (if applicable).
Evaluation of thyroid disorders | As clinically indicated
  blood draws, CT and other scans, physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Background] Klubo-Gwiezdzinska J, Wartofsky L. The Role of Molecular Diagnostics in the Management of Indeterminate Thyroid Nodules. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3507-3510. doi: 10.1210/jc.2018-01081. PMID 30032182
- [Background] Thakur S, Tobey A, Daley B, Auh S, Walter M, Patel D, Nilubol N, Kebebew E, Patel A, Jensen K, Vasko V, Klubo-Gwiezdzinska J. Limited Utility of Circulating Cell-Free DNA Integrity as a Diagnostic Tool for Differentiating Between Malignant and Benign Thyroid Nodules With Indeterminate Cytology (Bethesda Category III). Front Oncol. 2019 Sep 18;9:905. doi: 10.3389/fonc.2019.00905. eCollection 2019. PMID 31620364
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1977-DK-0096.html